CLINICAL TRIAL: NCT04424290
Title: A First-in Human Trial to Study Safety and Tolerability of Single Rising Intravitreal dOses (Open Label, Non-randomized, Uncontrolled) and in Addition the Early Biological Response of Multiple intravitReal Dosing (Single-masked, raNdomized, Sham-controlled) of BI 764524 in panretinaL Photocoagulation (PRP) Treated proLiferative Diabetic Retinopathy (PDR) Patients With Diabetic Macular Ischemia (DMI) - the HORNBILL Study
Brief Title: HORNBILL: A Study to Test Different Doses of BI 764524 in Patients Who Have Had Laser Treatment for a Type of Diabetic Eye Disease Called Diabetic Retinopathy With Diabetic Macular Ischemia
Acronym: HORNBILL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1436-0001; 2019-004432-28 (EudraCT Number)
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This trial will consist of an single rising dose (SRD) part followed by an multiple dosing (MD) part. SRD part will be nonrandomized, open-label, and uncontrolled. MD part will be single-masked, randomized and sham-controlled (Ratio 2:1). Parties masked in the MD part are participant and masked site staff (including investigator). The Intervention model in the MD part is active group versus sham injection (=2 arms).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single-rising dose part - low dose BI 764524 (Experimental): Pan-retinal photocoagulation (PRP)-treated proliferative diabetic retinopathy (PDR) patients with diabetic macular ischaemia (DMI) received one intravitreal injection of low dose BI 764524.
  Interventions: Drug: BI 764524
- Single-rising dose part - medium dose BI 764524 (Experimental): Pan-retinal photocoagulation (PRP)-treated proliferative diabetic retinopathy (PDR) patients with diabetic macular ischaemia (DMI) received one intravitreal injection of medium dose BI 764524.
  Interventions: Drug: BI 764524
- Single-rising dose part - high dose BI 764524 (Experimental): Pan-retinal photocoagulation (PRP)-treated proliferative diabetic retinopathy (PDR) patients with diabetic macular ischaemia (DMI) received one intravitreal injection of high dose BI 764524.
  Interventions: Drug: BI 764524
- Multiple dosing part - Sham (Sham Comparator): Pan-retinal photocoagulation (PRP)-treated proliferative diabetic retinopathy (PDR) patients with diabetic macular ischaemia (DMI) received three sham intravitreal injections, each separated by 4 weeks.
  Interventions: Drug: Sham control of BI 764524
- Multiple dosing part - high dose BI 764524 (Experimental): Pan-retinal photocoagulation (PRP)-treated proliferative diabetic retinopathy (PDR) patients with diabetic macular ischaemia (DMI) received three intravitreal injections of high dose BI 764524, each separated by 4 weeks.
  Interventions: Drug: BI 764524

INTERVENTIONS:
Drug: BI 764524 — BI 764524
  Arms: Multiple dosing part - high dose BI 764524; Single-rising dose part - high dose BI 764524; Single-rising dose part - low dose BI 764524; Single-rising dose part - medium dose BI 764524
Drug: Sham control of BI 764524 — Sham control of BI 764524
  Arms: Multiple dosing part - Sham

SUMMARY:
This is a study in people with a type of diabetic eye disease called diabetic retinopathy with diabetic macular ischemia. People who have had laser treatment for their diabetic retinopathy can participate in the study. The laser treatment is called panretinal photocoagulation.

The purpose of the study is to find out how well different doses of a medicine called BI 764524 are tolerated. BI 764524 is injected into the eye. The study has 2 parts. In the first part, participants get different doses of BI 764524 only once. Participants are in the first part for about 5 months and visit the study site about 8 times. In the second part, participants are put into different groups by chance. Some participants get BI 764524 injections every 4 weeks. Other participants get sham injections every 4 weeks. A sham injection means that it is not a real injection and contains no medicine. Participants cannot tell whether they get the real injection or a sham injection. For the second part, participants are in the study for about 7 months. During this time, they visit the study site about 7 times. In this study, BI 764524 is given to humans for the first time.

The doctors compare how well people tolerate the BI 764524 injections and the sham injections.

The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

Single rising dose (SRD) and multiple dosing (MD) part:

* Pan-retinal photo coagulation treated proliferative diabetic retinopathy (PDR) participants with either no or inactive retinal neovascularization per investigator judgement in the study eye
* Male or female participants of age ≥ 18 years
* HbA1c of ≤ 12.0%
* Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use two methods of contraception with at least one of them being a highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information and in the clinical trial protocol.

  --A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is NOT a method of permanent sterilisation. A postmenopausal state is defined as no menses for 2 years without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 2 years of menorrhea, a single FSH measurement is sufficient.
* Signed and dated written informed consent in accordance with ICH Harmonized Guideline for Good Clinical Practice (ICH GCP) and local legislation prior to admission to the trial

SRD part only:

* Evidence of diabetic macular ischemia (DMI) per investigator´s judgement, defined as any degree of disruption of retinal vascularity in superficial and/or deep retinal plexus in OCTA
* Best-corrected Visual activity (VA) in the non-study eye better than best-corrected VA in the study-eye, if both eyes are eligible and have identical VA the investigator may select the study eye.
* Best-corrected VA ≤55 letters (20/80) or worse

MD part only:

* Presence of significant DMI: large foveal avascular zone defined as those with ≥0.5mm2 area in superficial vascular complex (SVC) present on optical coherence tomography angiography. If FAZ is <0.5mm2 then enlarged peri-foveal inter-capillary space in at least 1 quadrant will be sufficient.
* If both eyes are eligible, the investigator may select either eye to be the study eye.
* Best-corrected VA ≤ 85 letters (20/20) or worse

Exclusion Criteria:

SRD part only:

* Participants receiving intravitreal (IVT) injections for active diabetic macular edema (DME, injections: anti-vascular endothelial growth factor (VEGF), steroids) and macular laser in the study eye in the previous 3 months prior to enrolment
* Participants receiving anti-VEGF IVT injections for active PDR in the study eye in the previous 3 months prior to enrolment
* Current or planned use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoximine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol)
* Additional eye disease in the study eye that could compromise best corrected VA (BCVA) with visual field loss, uncontrolled glaucoma (IOP>24), age related macular degeneration, history of ischemic optic neuropathy or retinal vascular occlusion, symptomatic vitreomacular traction, or genetic disorders such as retinitis pigmentosa; history of high myopia > 8 diopters in the study eye. Anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation with SD-OCT
* Any intraocular surgery in the study eye within 3 months prior to screening
* Aphakia or total absence of the posterior capsule. Yttrium aluminium garnet (YAG) laser capsulotomy in the study eye if performed less than 3 months prior to enrolment
* Participants not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator´s opinion, makes the patient an unreliable trial participant)
* Previous participation in this trial or in other trials with IVT injections administered within 3 months.

Further exclusion criteria apply.

MD part only:

* DME, defined as a central subfield thickness (CST) ≥305 micrometer (μm) for men and ≥290 μm women measured with optovue (Optical coherent tomography) OCT in the study eye
* Participants receiving IVT injections for active DME (anti-VEGF, steroids) and macular laser in the study eye in the previous 3 months prior to enrolment
* Participants receiving anti-VEGF IVT injections for active PDR in the study eye in the previous 3 months prior to enrolment
* Heavily lasered macula in the study eye per investigator's judgement
* History of vitrectomy in the study eye
* Epiretinal membrane with extended foveal contour distortion in the study eye per investigator's judgement
* Current or planned use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoximine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol) Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (13):
  - Trinity Research, Dothan, Alabama
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Stanford University Medical Center, Palo Alto, California
  - Florida Retina Institute, Orlando, Florida
  - Raj K. Maturi, MD PC, Carmel, Indiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Austin Research Center for Retina, PLLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
- United Kingdom (6):
  - Bradford Royal Infirmary, Bradford
  - Bristol Eye Hospital, Bristol
  - Southend University Hospital, Essex
  - Gloucestershire Royal Hospital, Gloucester
  - Moorfields Eye Hospital, London
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Chong V, Nguyen QD, Sepah Y, Giani A, Pearce E. HORNBILL: a phase I/IIa trial examining the safety, tolerability and early response of BI 764524 in patients with diabetic retinopathy and diabetic macular ischaemia-rationale, study design and protocol. Trials. 2022 Aug 17;23(1):669. doi: 10.1186/s13063-022-06527-y. PMID 35978329
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a trial consisting of a non-randomised, uncontrolled, open label single-rising dose part and a randomised, shamcontrolled, single-blind multiple dosing part.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Single-rising Dose Part - Low Dose BI 764524 | Single-rising Dose Part - Medium Dose BI 764524 | Single-rising Dose Part - High Dose BI 764524 | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Started | 3 | 3 | 7 | 10 | 22
Treated | 3 | 3 | 6 | 10 | 21
Completed | 3 | 3 | 6 | 7 | 20
Not Completed | 0 | 0 | 1 | 3 | 2
Not completed — Not treated | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Other than listed | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: all patients who were randomised and treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-rising Dose Part - Low Dose BI 764524 | Single-rising Dose Part - Medium Dose BI 764524 | Single-rising Dose Part - High Dose BI 764524 | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 10 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (15.0) | 61.0 (7.0) | 60.8 (6.0) | 60.0 (6.5) | 59.3 (13.2) | 60.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 5 | 10 | 21
  Male | 1 | 1 | 4 | 5 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 4 | 2 | 10
  Not Hispanic or Latino | 3 | 2 | 3 | 6 | 19 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 3 | 4
  White | 1 | 2 | 6 | 9 | 17 | 35
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Single-rising Dose (SRD) Part - The Number of Patients With Dose Limiting Events (DLEs) From Drug Administration Until Day 8
Description: Single-rising dose (SRD) part - The number of patients with dose limiting events (DLEs) from drug administration until Day 8 (7 days after treatment).
Time Frame: From drug administration (day 1) till day 8, Up to 7±2 days.
Population: Treated set: all patients who were randomised and treated with at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-rising Dose Part - Low Dose BI 764524 | Single-rising Dose Part - Medium Dose BI 764524 | Single-rising Dose Part - High Dose BI 764524
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 0

2. Primary Outcome: Multiple Dosing (MD) Part - the Number of Patients With Drug-related Adverse Events (AEs) From Drug Administration Until End of Trial.
Description: Multiple dosing (MD) part - the number of patients with drug-related Adverse Events (AEs) from drug administration until End of Trial.
Time Frame: From drug administration (day 1) till End of Trial, up to 23 weeks.
Population: Treated set: all patients who were randomised and treated with at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 10 | 21
Participants | 0 | 2

3. Secondary Outcome: SRD Part - Number of Patients With Drug-related Adverse Events at End of Trial
Description: SRD part - Number of patients with drug-related Adverse Events at End of Trial.
Time Frame: From drug administration (day 1) till End of Trial, up to 15 weeks.
Population: Treated set: all patients who were randomised and treated with at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-rising Dose Part - Low Dose BI 764524 | Single-rising Dose Part - Medium Dose BI 764524 | Single-rising Dose Part - High Dose BI 764524
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 0

4. Secondary Outcome: SRD Part - Number of Patients With Ocular Adverse Events (Eye Disorders) at End of Trial
Description: SRD part - Number of patients with ocular Adverse Events (eye disorders) at End of Trial.
Time Frame: From drug administration (day 1) till End of Trial, up to 15 weeks.
Population: Treated set: all patients who were randomised and treated with at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Single-rising Dose Part - Low Dose BI 764524 | Single-rising Dose Part - Medium Dose BI 764524 | Single-rising Dose Part - High Dose BI 764524
Number analyzed (Participants) | 3 | 3 | 6
Participants | 2 | 0 | 3

5. Secondary Outcome: MD Part - Number of Patients With Ocular Adverse Events (Eye Disorders) at End of Trial
Description: MD part - Number of patients with ocular Adverse Events (eye disorders) at End of Trial.
Time Frame: From drug administration (day 1) till End of Trial, up to 23 weeks.
Population: Treated set: all patients who were randomised and treated with at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 10 | 21
Participants | 4 | 4

6. Secondary Outcome: MD Part - Change From Baseline of the Size of the FAZ in FTR at Visit 5
Description: MD part - Change from baseline of the size of the foveal avascular zone (FAZ) in optical coherence tomography angiography (OCTA) in full thickness retina (FTR) at Visit 5. Results calculated as [Baseline data]-[Visit 5 data].
Time Frame: Baseline (day 0) and Visit 5 (day 85±7).
Population: All patients who were randomised and treated with at least one dose of study drug and with baseline and at least 1 on-treatment post-baseline value.
Measure: Mean (Standard Deviation); unit: Millimeter^2
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 7 | 16
Millimeter^2 | 0.0167 (0.0197) | -0.0004 (0.0381)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; The Mixed model with repeated measurements (MMRM) model included the fixed, categorical effects of treatment at each visit and the fixed continuous effects of baseline at each visit. Visit were treated as the repeated measure with an unstructured covariance structure used to model the within-patient measurements. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors; Test type: Other; Adjusted mean difference = -0.0234, 95% CI 2-sided [-0.0558 to 0.0089], Standard Error of Mean 0.0157 — Difference calculated as [BI]-[Sham]

7. Secondary Outcome: MD Part - Change From Baseline of the Size of the FAZ in SVC at Visit 5
Description: MD part - Change from baseline of the size of the foveal avascular zone (FAZ) in optical coherence tomography angiography (OCTA) in superficial vascular complex (SVC) at Visit 5. Results calculated as [Baseline data]-[Visit 5 data].
Time Frame: Baseline (day 0) and Visit 5 (day 85±7).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter^2
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 8 | 15
Millimeter^2 | 0.0489 (0.0740) | 0.0741 (0.1130)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = 0.0215, 95% CI 2-sided [-0.0670 to 0.1100], Standard Error of Mean 0.0429 — Difference calculated as [BI]-[Sham]

8. Secondary Outcome: MD Part - Change From Baseline of the Size of the FAZ in FTR at Visit 7
Description: MD part - Change from baseline of the size of the foveal avascular zone (FAZ) in optical coherence tomography angiography (OCTA) in full thickness retina (FTR) at Visit 7. Results calculated as [Baseline data]-[Visit 7 data].
Time Frame: Baseline (day 0) and Visit 7 (day 155±7).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter^2
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 7 | 16
Millimeter^2 | 0.0133 (0.0152) | -0.0027 (0.0345)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = -0.0109, 95% CI 2-sided [-0.0412 to 0.0195], Standard Error of Mean 0.0145 — Difference calculated as [BI]-[Sham]

9. Secondary Outcome: MD Part - Change From Baseline of the Size of the FAZ in SVC at Visit 7
Description: MD part - Change from baseline of the size of the foveal avascular zone (FAZ) in optical coherence tomography angiography (OCTA) in superficial vascular complex (SVC) at Visit 7. Results calculated as [Baseline data]-[Visit 7 data].
Time Frame: Baseline (day 0) and Visit 7 (day 155±7).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter^2
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 7 | 14
Millimeter^2 | 0.1233 (0.1473) | 0.1101 (0.1445)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = -0.0228, 95% CI 2-sided [-0.1477 to 0.1021], Standard Error of Mean 0.0603 — Difference calculated as [BI]-[Sham]

10. Secondary Outcome: MD Part - Change From Baseline of Best Corrected Visual Acuity (BCVA) at Visit 3
Description: Change from baseline of best corrected visual acuity (BCVA) at Visit 3. BCVA was measured using the early treatment diabetic retinopathy study (ETDRS) visual acuity (VA) chart starting at a test distance of 4 meter. The BCVA score was the number of letters read correctly by the patient. Results calculated as [Baseline data]-[Visit 3 data].
Time Frame: Baseline (day 0) and Visit 3 (day 29±7).
Population: All patients who were randomised and treated with at least one dose of study drug, with data for the baseline and the corresponding visit.
Measure: Mean (Standard Deviation); unit: Number of letters
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 10 | 20
Number of letters | 1.5 (13.5) | 1.1 (5.2)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = -1.3, 95% CI 2-sided [-8.1 to 5.5], Standard Error of Mean 3.3 — Difference calculated as [BI]-[Sham]

11. Secondary Outcome: MD Part - Change From Baseline of Best Corrected Visual Acuity (BCVA) at Visit 4
Description: Change from baseline of best corrected visual acuity (BCVA) at Visit 4. BCVA was measured using the early treatment diabetic retinopathy study (ETDRS) visual acuity (VA) chart starting at a test distance of 4 meter. The BCVA score was the number of letters read correctly by the patient. Results calculated as [Baseline data]-[Visit 4 data].
Time Frame: Baseline (day 0) and Visit 4 (day 57±7).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Number of letters
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 10 | 20
Number of letters | -4.1 (24.4) | 1.4 (6.0)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = 4.4, 95% CI 2-sided [-7.3 to 16.2], Standard Error of Mean 5.7 — Difference calculated as [BI]-[Sham]

12. Secondary Outcome: MD Part - Change From Baseline of Best Corrected Visual Acuity (BCVA) at Visit 5
Description: Change from baseline of best corrected visual acuity (BCVA) at Visit 5. BCVA was measured using the early treatment diabetic retinopathy study (ETDRS) visual acuity (VA) chart starting at a test distance of 5 meter. The BCVA score was the number of letters read correctly by the patient. Results calculated as [Baseline data]-[Visit 5 data].
Time Frame: Baseline (day 0) and Visit 5 (day 85±7).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Number of letters
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 10 | 17
Number of letters | 3.9 (10.7) | 2.5 (6.5)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = -3.3, 95% CI 2-sided [-9.6 to 3.0], Standard Error of Mean 3.1 — Difference calculated as [BI]-[Sham]

13. Secondary Outcome: MD Part - Change From Baseline of Best Corrected Visual Acuity (BCVA) at Visit 6
Description: Change from baseline of best corrected visual acuity (BCVA) at Visit 6. BCVA was measured using the early treatment diabetic retinopathy study (ETDRS) visual acuity (VA) chart starting at a test distance of 6 meter. The BCVA score was the number of letters read correctly by the patient. Results calculated as [Baseline data]-[Visit 6 data].
Time Frame: Baseline (day 0) and Visit 6 (day 113±7).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Number of letters
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 10 | 17
Number of letters | 2.6 (9.6) | 3.1 (9.8)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = -0.6, 95% CI 2-sided [-7.3 to 6.1], Standard Error of Mean 3.3 — Difference calculated as [BI]-[Sham]

14. Secondary Outcome: MD Part - Change From Baseline of Best Corrected Visual Acuity (BCVA) at Visit 7
Description: Change from baseline of best corrected visual acuity (BCVA) at Visit 7. BCVA was measured using the early treatment diabetic retinopathy study (ETDRS) visual acuity (VA) chart starting at a test distance of 7 meter. The BCVA score was the number of letters read correctly by the patient. Results calculated as [Baseline data]-[Visit 7 data].
Time Frame: Baseline (day 0) and Visit 7 (day 155±7).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Number of letters
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 10 | 19
Number of letters | 4.9 (9.3) | 3.4 (7.5)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = -2.8, 95% CI 2-sided [-8.7 to 3.1], Standard Error of Mean 2.9 — Difference calculated as [BI]-[Sham]

15. Secondary Outcome: MD Part - Change From Baseline of Central Retinal Thickness (CRT) at Visit 3
Description: MD part - Change from baseline of central retinal thickness (CRT) in Spectral domain optical coherence tomography (SD-OCT) at Visit 3. Results calculated as [Baseline data]-[Visit 3 data].
Time Frame: Baseline (day 0) and Visit 3 (day 29±7).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Micrometer
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 10 | 20
Micrometer | 1.6 (4.9) | 0.9 (7.2)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = 0.2, 95% CI 2-sided [-4.9 to 5.4], Standard Error of Mean 2.5 — Difference calculated as [BI]-[Sham]

16. Secondary Outcome: MD Part - Change From Baseline of Central Retinal Thickness (CRT) at Visit 4
Description: MD part - Change from baseline of central retinal thickness (CRT) in Spectral domain optical coherence tomography (SD-OCT) at Visit 4. Results calculated as [Baseline data]-[Visit 4 data].
Time Frame: Baseline (day 0) and Visit 4 (day 57±7)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Micrometer
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 9 | 19
Micrometer | -1.7 (5.1) | 0.2 (7.2)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = 2.6, 95% CI 2-sided [-2.7 to 7.9], Standard Error of Mean 2.6 — Difference calculated as [BI]-[Sham]

17. Secondary Outcome: MD Part - Change From Baseline of Central Retinal Thickness (CRT) at Visit 5
Description: MD part - Change from baseline of central retinal thickness (CRT) in Spectral domain optical coherence tomography (SD-OCT) at Visit 5. Results calculated as [Baseline data]-[Visit 5 data].
Time Frame: Baseline (day 0) and Visit 5 (day 85±7).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Micrometer
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 9 | 17
Micrometer | -2.9 (5.3) | 3.9 (12.8)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = 7.7, 95% CI 2-sided [-1.2 to 16.5], Standard Error of Mean 4.3 — Difference calculated as [BI]-[Sham]

18. Secondary Outcome: MD Part - Change From Baseline of Central Retinal Thickness (CRT) at Visit 6
Description: MD part - Change from baseline of central retinal thickness (CRT) in Spectral domain optical coherence tomography (SD-OCT) at Visit 6. Results calculated as [Baseline data]-[Visit 6 data].
Time Frame: Baseline (day 0) and Visit 6 (day 113±7).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Micrometer
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 9 | 17
Micrometer | -3.0 (3.8) | 8.6 (25.1)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = 13.8, 95% CI 2-sided [-2.3 to 29.8], Standard Error of Mean 7.8 — Difference calculated as [BI]-[Sham]

19. Secondary Outcome: MD Part - Change From Baseline of Central Retinal Thickness (CRT) at Visit 7
Description: MD part - Change from baseline of central retinal thickness (CRT) in Spectral domain optical coherence tomography (SD-OCT) at Visit 7. Results calculated as [Baseline data]-[Visit 7 data].
Time Frame: Baseline (day 0) and Visit 7 (day 155±7).
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Micrometer
Arm/Group | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
Number analyzed (Participants) | 9 | 19
Micrometer | -3.2 (7.4) | 3.5 (9.5)
Statistical Analysis 1: Comparison: Multiple Dosing Part - Sham vs Multiple Dosing Part - High Dose BI 764524; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted mean difference = 6.8, 95% CI 2-sided [-0.9 to 14.5], Standard Error of Mean 3.7 — Difference calculated as [BI]-[Sham]

ADVERSE EVENTS:
Time Frame: From time of administration till the End of Trial, up to 15 weeks for the SRD part and up to 23 weeks for the MD part.
Description: Treated set: all patients who were randomised and treated with at least one dose of study drug.
Arm/Group | Single-rising Dose Part - Low Dose BI 764524 | Single-rising Dose Part - Medium Dose BI 764524 | Single-rising Dose Part - High Dose BI 764524 | Multiple Dosing Part - Sham | Multiple Dosing Part - High Dose BI 764524
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/10 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/6 | 3/10 | 2/21
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 5/6 | 6/10 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-rising Dose Part - Low Dose BI 764524 (N=3) | Single-rising Dose Part - Medium Dose BI 764524 (N=3) | Single-rising Dose Part - High Dose BI 764524 (N=6) | Multiple Dosing Part - Sham (N=10) | Multiple Dosing Part - High Dose BI 764524 (N=21)
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 2 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-rising Dose Part - Low Dose BI 764524 (N=3) | Single-rising Dose Part - Medium Dose BI 764524 (N=3) | Single-rising Dose Part - High Dose BI 764524 (N=6) | Multiple Dosing Part - Sham (N=10) | Multiple Dosing Part - High Dose BI 764524 (N=21)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 1 | 0
Episcleritis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Iris neovascularisation (Eye disorders) | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vitreal cells (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 2 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood folate increased (Investigations) | 0 | 0 | 0 | 0 | 2
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 0 | 0 | 2 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT04424290/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT04424290/SAP_001.pdf